CLINICAL TRIAL: NCT01357902
Title: An Open Label, Randomized, Cross-Over Study to Investigate the Single Dose Bioequivalence of Lamotrigine Dispersible/Chewable Tablets (5mg) Compared to Lamotrigine Compressed/Standard Tablets (25mg) in Chinese Healthy Male Subjects
Brief Title: Lamotrigine Bioequivalence Study to Compare Dispersible Tables With Compressed Tablets in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115261
Record Dates: First submitted 2011-05-12; First posted 2011-05-23 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

ARMS (1):
- Lamictal (Experimental): Chinese healthy male subjects were randomized to receive single dose of either 5 mg lamotrigine dispersible/chewable tablets or 25mg compressed/standard tablets.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine is a selective inhibitor of a voltage-sensitive sodium channel, is an anti-epileptic drug of the phenyltriazine class.

SUMMARY:
It is an open-label, randomised, single dose, two-sequence cross-over study. Twenty-four eligible, healthy, Chinese male subjects will be enrolled after providing written informed consent. Subjects will be randomised into two treatment groups 1 day prior to the first dosing day and will be assigned to regimen sequences (AB or BA) in a balanced fashion in accordance with the randomisation schedule. Regimen A is five lamotrigine 5 mg chewable/dispersible tablets and Regimen B is one lamotrigine 25 mg standard/compressed tablet.

Subjects will receive their allocated regimen on the morning of Day 1 and will undergo study assessments for 7 days (until Day 8). Subjects will receive their alternate randomised treatment after a washout period of 14-21 days from Day 1. Subjects will undergo a further assessment period of 7 days and will attend a follow-up visit during 8-12 days after the second treatment. The total observation period in this study will be 23~34 days.

Subjects will arrive at the research unit on the evening before each lamotrigine dosing occasion and will remain in the unit until the 24-h post-dose evaluations have been completed (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 h). After this, subjects will return home but must return to the unit for further assessments to be made at 36, 48, 72, 96, 120, 144 and 168 h after dosing Study Endpoints/Assessments A total of 19 serial blood samples (5 mL each) will be collected for the measurement of plasma lamotrigine concentrations at each study assessment. Safety and tolerability assessments (monitoring of adverse events and serious adverse events, routine laboratory determinations, vital sign measurements and 12-lead electrocardiogram) will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. According to medical history and clinical examination, healthy and non-smoking male subjects
2. Between 18 and 45 years of age, inclusive.
3. Body weight >=50 kg and BMI 19-24 kg/m2, inclusive.
4. Male subjects with female partners of child-bearing potential must agree to use one of the following contraceptive methods after the first dose of study treatment and until the follow up visit:

   * Condom plus partner use of a highly effective contraceptive such as occlusive cap (diaphragm or cervical/vault cap) plus spermicidal agent (foam/gel/film/cream/suppository), oral contraceptive, injectable progesterone, implant of etonogestrel or levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, or intrauterine device. OR,
   * Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
5. Good compliance with research policies, procedures and restrictions.
6. Can read and understand the informed consent. Informed consent should be obtained prior to admission to the study.
7. No abnormality revealed by the laboratory tests, or any slight abnormality judged by the investigator to have no clinical significance.
8. Aspartate aminotransferase (AST), ALT, alkaline phosphatase and bilirubin=<1.5 x upper limit of normal (ULN).
9. Normal systolic (90-140 mmHg) and diastolic (<90 mmHg) blood pressure at screening, and normal pulse (supine).
10. A normal 12-lead ECG at pre-study screening.
11. Single or average QT duration corrected for heart rate by Bazett's formula (QTcB) or by Fridericia's formula (QTcF) <450 msec; or QTc <480 msec in subjects with bundle branch block.
12. Liver serum virological and human immunodeficiency virus tests are negative

Exclusion Criteria:

1. Any clinically relevant abnormality identified on the screening history and physical or laboratory examination significant cardiovascular, neurological, psychiatric, haematological or renal abnormalities.
2. Definite or suspected personal history or family history of adverse reactions or hypersensitivity to the study drug or to drugs with a similar chemical structure.
3. Participation in a clinical trial within the 30 days before the start of the study.
4. The subject has received prescribed medication or over-the-counter (OTC) medicine including herbal medicines within 14 days before the first dosing day. The use of lubricant with spermicide or contraceptive barrier devices and other contraceptives is permitted.
5. History of any clinically significant illness within 4 weeks before the study.
6. History of any clinically significant physical or organic abnormalities.
7. Abnormalities of 12-lead ECG which the investigators think increase the risk of participation in the study.
8. History of liver dysfunction such as jaundice, or hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCAb) positive regardless of ALT level or ALT greater than or equal to 2-times ULN. Subjects with Gilbert's syndrome will be excluded from the study.
9. Positive pre-study screening result for hepatitis B antigen, hepatitis C antibodies or HIV-1 or HIV-2 antibody.
10. Subject whose HLA-B*1502 is positive will be exclude from the study.
11. Abuse of alcohol, defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units. One unit is equivalent to half a pint (~ 240 mL) of beer, one (25 mL) measure of spirits or one glass (125 mL) of wine.
12. Positive pre-study drug/alcohol screen.
13. History of obvious active haematological disorder or significant blood loss in the past 3 months.
14. Subject donated blood within a 56-day period or donated plasma within 1 week prior the study.
15. Subject is mentally or legally incapacitated.
16. Any other reason at the Investigators' discretion

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04-18 (Actual); Primary Completion 2011-05-23 (Actual); Study Completion 2011-05-23 (Actual)

PRIMARY OUTCOMES:
AUC(0-infinity) | taken pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h after each dosing
AUC(0-t) | taken pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h after each dosing
Cmax | taken pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h after each dosing

SECONDARY OUTCOMES:
tmax | taken pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h after each dosing
terminal phase half-life | taken pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h after each dosing
12-lead electrocardiogram (ECG), vital signs, nursing observations, spontaneous adverse experience reporting and laboratory safety data | at Screening, Day 0, Day1-8, Day15-22 and follow up 7-14 days after second dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shatin, New Territories, Hong Kong

REFERENCES:
- See also: Results for study 115261 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115261?search=study&search_terms=115261#rs